CLINICAL TRIAL: NCT00176878
Title: Bone Marrow Transplantation for Non-Malignant Congenital Bone Marrow Failure Disorders
Brief Title: Stem Cell Transplant for Bone Marrow Failure Syndromes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT2000-18; 9504M09637 (Other: IRB, University of Minnesota); NCT00005895 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-08-06 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Diamond-Blackfan Anemia; Kostmann's Neutropenia; Shwachman-Diamond Syndrome
Keywords: Stem cell transplant; T-cell depletion; TLI; bone marrow failure disorders
MeSH Terms: conditions — Anemia, Diamond-Blackfan; Shwachman-Diamond Syndrome; Bone Marrow Failure Disorders | interventions — Stem Cell Transplantation; fludarabine phosphate; Busulfan; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone Marrow Failure Disorders (Experimental): Patients with Diamond-Blackfan Anemia, Kostmann's Neutropenia, Shwachman-Diamond Syndrome
  Interventions: Procedure: Stem cell transplant; Drug: Fludarabine monophosphate; Procedure: Total lymphoid irradiation; Drug: Busulfan; Biological: anti-thymocyte globulin

INTERVENTIONS:
Procedure: Stem cell transplant — Stem cell transplant on Day 0 - healthy marrow from an unrelated individual. A minimum of 1.0 x 10^9/kg nucleated cells/kg ideal body weight will be collected with a goal of 2.0 x 10^9/kg.
  Other Names: BMT
Drug: Fludarabine monophosphate — fludarabine 175 mg/m^2 (total) on Days -6 through -3.
  Other Names: Fludara
Procedure: Total lymphoid irradiation — Dose 500 cGy radiation therapy to specific areas of the body
  Other Names: TLI
Drug: Busulfan — Busulfan 8 mg/kg (total) on Days - 8 and -7 (orally or through the catheter),
  Other Names: Busulfex
Biological: anti-thymocyte globulin — anti-thymocyte globulin (ATG) 15 mg/kg on days -2 and -1 via catheter
  Other Names: ATG

SUMMARY:
The researchers hypothesize that it will be possible to perform unrelated bone marrow or cord blood transplants in a safer manner by using less intensive therapy yet still achieve an acceptable level of donor cell engraftment for non-malignant congenital bone marrow failure disorders.

DETAILED DESCRIPTION:
Prior to transplantation, subjects will receive the drugs busulfan (orally or through the catheter), as well as fludarabine and anti-thymocyte globulin (ATG) via the catheter. Busulfan, fludarabine and ATG will be given with Total Lymphoid Irradiation (TLI) to help the new donor bone marrow take and grow after transplantation.

Those patients receiving donor marrow will have the T cells (a type of white blood cell in the donor marrow) removed to lower the risk that the new marrow will react to their body, a condition called Graft-Versus-Host-Disease (GVHD). After bone marrow transplantation, subjects will receive drugs to help prevent GVHD, including cyclosporin and mycophenolate mofetil (MMF).

Blood samples are taken at day 28, day 60, day 100, 1 year and as required by medical status yearly for five years after transplant to evaluate how well the new marrow is growing. A bone marrow biopsy is required at day 21, at day 100 and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for transplantation under this protocol will be <35 years of age, and will be diagnosed with:

  * a bone marrow failure syndrome unresponsive to available therapy, including but not limited to Diamond-Blackfan anemia, Shwachman Diamond syndrome or Kostmann's neutropenia but exclusive of aplastic anemia.
* Diamond Blackfan Anemia:

  * Patients must show evidence of steroid resistance requiring equivalent of >6 transfusions yearly despite steroid therapy.
  * Evidence of developing aplasia or myelodysplasia will also be criteria for transplantation.
* Kostmann's Neutropenia, Shwachman-Diamond syndrome:

  * Patients must have been previously diagnosed as having a clinical picture characteristic of Shwachman-Diamond syndrome (exocrine pancreatic insufficiency, growth retardation, metaphyseal dysostosis, neutropenia), or must have a bone marrow aspirate consistent with Kostmann's neutropenia, with no evidence of acute leukemia.
  * Patients must have failed therapy with granulocyte-colony stimulating factor (G-CSF), as determined by an inability to maintain an absolute neutrophil count (ANC) >750 cells/ml(3), or manifesting recurrent infections despite G-CSF administration resulting in life threatening infections or repeated hospitalizations (<4 /year).

Exclusion Criteria:

* Patients >35 years of age
* Karnofsky score <70%
* Hepatic dysfunction as determined by bilirubin >3.0, ALT >150, or active hepatitis
* Pulmonary function tests with forced volume vital capacity (FVC) and forced expiratory volume (FEV) <70%; O2 saturation <94%
* Renal dysfunction with glomerular filtration rate (GFR) <30% of predicted.
* Cardiac compromise, with left ejection fraction <45%.
* Severe, stable neurologic impairment.
* Human immunodeficiency virus (HIV) positivity.
* Pregnant or lactating females

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2000-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — University of Minnesota Medical Center
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow Failure Patients: All patients with non-malignant, congenital bone marrow failure disorders and treated with stem cell transplant, chemotherapy (Busulfan, ATG, Fludarabine) and irradiation.
Period: Overall Study
Arm/Group | Bone Marrow Failure Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bone Marrow Failure Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive (Survival) at 2 Years
Description: Calculated from day 1 of transplant to last contact.
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | Bone Marrow Failure Patients
Number analyzed (Participants) | 10
Participants | 6

2. Secondary Outcome: Number of Patients Alive at Three Years (Survival)
Description: Number of subjects who survived 3 years post-transplant.
Time Frame: 3 years
Measure: Number; unit: Participants
Arm/Group | Bone Marrow Failure Patients
Number analyzed (Participants) | 10
Participants | 6

3. Secondary Outcome: Number of Patients With Succcessful Engraftment After Transplantation
Description: Number of patients who received non-genotypic identical marrow or cord blood cells using a "non-myeloablative" preparative regimen and exhibited engraftment at Day 42.
Time Frame: 42 Days
Measure: Number; unit: Participants
Arm/Group | Bone Marrow Failure Patients
Number analyzed (Participants) | 10
Participants | 10

4. Secondary Outcome: Number of Patients With Grade 2-4 Acute Graft Versus Host Disease
Description: Number of patients with Grade 2, 3 and 4 Acute (normally observed within the first 100 days) Graft Versus Host Disease. Acute GVHD is staged as follows: overall grade (skin-liver-gut) with each organ staged individually from a low of 1 to a high of 4. Patients with grade IV GVHD usually have a poor prognosis. Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening.
Time Frame: 100 Days
Measure: Number; unit: Participants
Arm/Group | Bone Marrow Failure Patients
Number analyzed (Participants) | 10
Participants | 5

5. Secondary Outcome: Number of Patients With Chronic Graft Versus Host Disease
Description: Number of patients who exhibited chronic (normally occurs after 100 days) Graft Versus Host Disease at 2 years post transplant. Chronic graft-versus-host-disease, over its long-term course, can also cause damage to the connective tissue and exocrine glands.
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | Bone Marrow Failure Patients
Number analyzed (Participants) | 10
Participants | 3

6. Secondary Outcome: Number of Patients With Disease Recurrence
Description: Number of patients who exhibited disease recurrence at 2 years.
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | Bone Marrow Failure Patients
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: Day 1 of study up through 1 year
Description: Only serious adverse events are reported. Other adverse events were not collected.
Arm/Group | Bone Marrow Failure Patients
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Failure Patients (N=10)
Bone marrow graft failure (Blood and lymphatic system disorders) | 3 (3) — Autologous recovery, Chimerism (secondary)
Death (General disorders) | 3 (3)
Graft-versus-host disease (acute) (Blood and lymphatic system disorders) | 1 (1) — Grade III-IV

LIMITATIONS AND CAVEATS:
Pharmacokinetic parameters in patients receiving 2 mg/kg/dose of busulfan twice daily was not performed. No data is available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes